CLINICAL TRIAL: NCT03449602
Title: A Randomized Trial Comparing the Diagnostic Sensitivity and Safety of Mini-thoracoscopy Versus Conventional Rigid Thoracoscopy in Undiagnosed Pleural Effusions
Brief Title: Minirigid Versus Conventional Rigid Thoracoscopy in Undiagnosed Pleural Effusions
Acronym: MICRO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Sahajal Dhooria, Assistant Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: NK/3695/Res
Record Dates: First submitted 2018-02-17; First posted 2018-02-28 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Pleural Effusion
Keywords: thoracoscopy; pleuroscopy; metastatic cancer; lung cancer; malignant pleural effusion; tuberculosis
MeSH Terms: conditions — Pleural Effusion; Neoplasm Metastasis; Lung Neoplasms; Pleural Effusion, Malignant; Tuberculosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mini-thoraoscopy (Experimental): The mini-thoracoscope manufactured by Richard Wolf GmbH, Knettligen, Germany will be used for performing thoracoscopic pleural biopsies. It has an outer diameter of 5.5 mm and a working channel diameter of 3.5 mm.
  Interventions: Device: Mini-thoracoscopy
- Conventional rigid thoracoscopy (Active Comparator): The rigid thoracoscope manufactured by Richard Wolf GmbH, Knettligen, Germany will be used for performing thoracoscopic pleural biopsies. It has an outer diameter of 10 mm and channel internal diameter of 5 mm.
  Interventions: Device: Conventional rigid thoraoscopy

INTERVENTIONS:
Device: Mini-thoracoscopy — Thoracoscopic pleural biopsy with the mini-thoracoscope
  Arms: Mini-thoraoscopy
Device: Conventional rigid thoraoscopy — Thoracoscopic pleural biopsy with the conventional rigid thoraoscope
  Arms: Conventional rigid thoracoscopy

SUMMARY:
Consecutive patients who are planned to undergo a medical thoracoscopy for obtaining pleural biopsies will be enrolled in the study.

One hundred subjects will be randomized in 1:1 ratio to undergo thoracoscopy to the following groups:

Group A (mini-thoracoscopy) Group B (Conventional rigid thoracoscopy) Primary outcome: (a) diagnostic sensitivity of mini-thoracoscopy and conventional rigid thoracoscopy in the diagnosis of exudative pleural effusions

DETAILED DESCRIPTION:
A significant proportion of patients with pleural effusions remain undiagnosed after performance of diagnostic procedures including cytological and microbiologic analysis of the pleural fluid and closed pleural biopsies. In this study, the investigators plan to compare the yield and safety of mini-thoracoscopy and conventional rigid thoracoscopy with the larger diameter scope.

This is a prospective study that will be conducted at the Thoracic Endoscopy Suite of the Department of Pulmonary Medicine, PGIMER, Chandigarh.

Consecutive patients who are planned to undergo a medical thoracoscopy for obtaining pleural biopsies will be enrolled in the study

One hundred subjects will be randomized in 1:1 ratio to undergo thoracoscopy. The randomization sequence will be generated using a computer (in blocks of 10), and the allocation will be placed in opaque sealed envelopes. The patients will be randomized to the following groups:

Group A (mini-thoracoscopy): The mini-thoracoscope manufactured by Richard Wolf GmbH, Knettligen, Germany will be used. It has an outer diameter of 5.5 mm and a working channel diameter of 3.5 mm.

Group B (Conventional rigid thoracoscopy): The rigid thoracoscope manufactured by Richard Wolf GmbH, Knettligen, Germany will be used that has an outer diameter of 10 mm and channel internal diameter of 5 mm.

Primary outcome: (a) diagnostic sensitivity of mini-thoracoscopy and conventional rigid thoracoscopy in the diagnosis of exudative pleural effusions.

ELIGIBILITY:
Inclusion Criteria:

* Medical thoracoscopy being performed for obtaining a pleural biopsy

Exclusion Criteria:

* PaO2/FIO2< 300; Hemodynamic instability Myocardial infarction or unstable angina in the last 6 wk Lack of pleural space due to adhesions Uncorrected coagulopathy Failure to provide informed consent

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Diagnostic sensitivity (intention-to-treat) | 6 months
  Difference between the diagnostic sensitivity of mini-thoracoscopy and conventional rigid thoracoscopy in the diagnosis of exudative pleural effusions by calculating the number of true positives diagnosed by thoracoscopic biopsy in the two groups out of the total diseased
Diagnostic sensitivity (per protocol) | 6 months
  Diagnostic sensitivity of mini-thoracoscopy and conventional rigid thoracoscopy in the diagnosis of exudative pleural effusions by calculating the number of true positives diagnosed by thoracocopic biopsy. In this analysis, the subjects crossed over to the rigid group (due to failure of minirigid to yield biopsy tissue) will be considered in the rigid group

SECONDARY OUTCOMES:
Sedative and analgesic dose | 1 day
  Comparing doses of sedative and analgesic agents required in the two groups
Pain scores by visual analog scale | 1 day
  Difference between intraoperative pain score associated with the use of the two devices (assessed after the procedure using the visual analog scale from 0-no pain to 100-maximum possible pain) in the two groups
Diagnostic specificity | 6 months
  Difference between the diagnostic specificity of mini-thoracoscopy and conventional rigid thoracoscopy in the diagnosis of exudative pleural effusions by calculating the number of true negatives diagnosed by thoracoscopic biopsy in the two groups out of those not diseased
Adverse effects | 1 month
  Differences between number of participants with treatment-related adverse events as assessed by CTCAE v4.0 in the two groups
Scope maneuverability | 1 day
  Differences between maneuverability of the two thoracoscopes on a visual analog scale (0-100 mm) assessed by the operator
Ease of obtaining biopsy | 1 day
  Differences between ease of obtaining pleural biopsy with the two thoracoscopes on a visual analog scale (0-100 mm) assessed by the operator
Incision size | 1 day
  Difference in the size of the incision required with the use of the two devices
Procedure duration | 1 day
  Difference in the duration of procedure in the two groups
Pain scores by Wong Baker FACES pain rating scale | 1 day
  Difference between intraoperative pain score associated with the use of the two devices (assessed after the procedure using the Wong Baker FACES pain rating scale) in the two groups

CONTACTS AND LOCATIONS:
Locations (1):
- Postgraduate Institute of Medical Education and Research, Chandigarh, India